CLINICAL TRIAL: NCT02493959
Title: Degradation of the Anorexic Hormone Peptide YY
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Hvidovre University Hospital (Other)
Collaborators: University of Copenhagen (Other)
Responsible Party: Principal Investigator, Kirstine Nyvold Bojsen-Moeller, MD, Hvidovre University Hospital
Allocation: Not Applicable | Model: Single Group | Masking: Single | Purpose: Basic Science
Other Study IDs: STKBM-PI14
Record Dates: First submitted 2015-07-02; First posted 2015-07-10 (Estimated); Last update posted 2015-07-10 (Estimated); Status verified 2015-07

CONDITIONS: Healthy
Keywords: PYY; Degradation; kinetics; men
MeSH Terms: conditions — Multiple Endocrine Neoplasia Type 1 | interventions — Sitagliptin Phosphate

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- PYY infusion (Experimental): IV infusion on 4 separate days of PYY or saline in Healthy, normal-weight men, age 18-50 years
  Interventions: Biological: PYY1-36 infusion; Biological: PYY1-36 + sitagliptin; Biological: PYY3-36 infusion; Biological: placebo

INTERVENTIONS:
Biological: PYY1-36 infusion — Infusion of 1.6 pmol/kg/min PYY1-36 for 2 hrs.
Biological: PYY1-36 + sitagliptin — Infusion of 1.6 pmol/kg/min PYY1-36 for 2 hrs. Two doses of 100 mg sitagliptin are administered 10 and 1 hour before start of infusion, respectively.
Biological: PYY3-36 infusion — 0.8 pmol/kg/min infusion of PYY3-36.
Biological: placebo — Infusion of saline for 2 hrs.

SUMMARY:
Peptide YY (PYY) is a gastrointestinal hormone released from the enteroendocrine cell upon food intake. The N-terminal truncated form, PYY3-36, exerts anorexic effects. In this study we want to investigate the kinetics of PYY1-36 and PYY3-36 and to examine whether a C-terminally degraded metabolite, PYY3-34, is formed after infusion of PYY.

ELIGIBILITY:
Inclusion Criteria:

* Healthy
* Normal BMI (18.5-25kg/m2)

Exclusion Criteria:

* Diabetes Mellitus
* Gastric bypass
* Non-caucasian
* Height changes >3 kg within last two months
* Hemoglobin < 7.6 mmol/l
* Chronic disease
* Smoking
* Regularly use of medicine
* Drug abuse

Ages: 18 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 8 (Actual)
Dates: Start 2014-05; Primary Completion 2015-07 (Actual); Study Completion 2015-07 (Actual)

PRIMARY OUTCOMES:
PYY3-34 concentration | 0-240 min
Half-lives of PYY1-36 and PYY3-36 | 0-240 min

OTHER OUTCOMES:
Appetite and nausea scores | 0-240 min
  Between infusion differences in VAS scores
Blood pressure | 0-240 min
  Between infusion differences in blood pressure
Blood glucose | 0-240 min
  Between infusion differences in blood glucose
Heart rate | 0-240 min
  Between infusion differences in heart rate

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Endocrinology, Hvidovre Hospital, Hvidovre, Denmark